CLINICAL TRIAL: NCT00672672
Title: Autologous Platelet Gel in Wound Healing of Coronary Artery Bypass Grafting (CABG) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed with no subjects accrued. PI decided to stop study.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0065-08-FB
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Wounds; Infection
Keywords: surgical site healing treated with autologous platlet gel
MeSH Terms: conditions — Wounds and Injuries; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Gel (Experimental): Participants receive platlet gel.
  Interventions: Biological: autologous platelet gel
- Control (No platelet gel) (Placebo Comparator): Participants do not receive platlet gel.
  Interventions: Biological: autologous platelet gel

INTERVENTIONS:
Biological: autologous platelet gel — Patients will receive APG to the surgical site in the operating room. The control site will receive no treatment.

SUMMARY:
This study will determine if autologous platelet gel (APG) on sternal incision and conduit sites will improve wound healing and decrease infection in coronary artery bypass grafting surgery patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the use of autologous platelet gel (APG) on sternal incision and conduit sites will improve wound healing and decrease the incidence of infection in patients undergoing coronary artery bypass grafting surgery

ELIGIBILITY:
Inclusion Criteria:

* Any patient who meets criteria and consents to undergo a CABG procedure involving conduit sites and consents to this study.

Exclusion Criteria:

* Any patient, after inclusion, whom is later determined to have had on-going therapy that could influence wound healing such as radiation or chemotherapy, extensive steroid use, or accidental trauma such as burns, etc.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01-13 (Actual); Primary Completion 2010-01-06 (Actual); Study Completion 2010-01-06 (Actual)

PRIMARY OUTCOMES:
Healing and infection of surgical sites | 30 days
  The surgical sites will be assessed for degree of healing and signs and symptoms of infection on post-op days one and three and during the patients' follow up visits in the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khoynezhad, MD, Principal Investigator — University of Nebraska